CLINICAL TRIAL: NCT01515241
Title: EXPLORATORY STUDY OF PLAQUE REGRESSION:A Phase II Single Center Open-Label Exploratory Trial of the Effect of CER 001 in Subjects With Familial Hypercholesterolemia
Brief Title: Exploratory Study of Plaque Regression
Acronym: EXPRESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cerenis Therapeutics, SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CER-001-CLIN-005
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-01

CONDITIONS: Heterozygous Familial Hypercholesterolemia
Keywords: Heterozygous Familial Hypercholesterolemia; Familial Hypercholesterolemia; HDL mimetic; ApoA-1
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — CER-001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label single arm study of CER-001 (Other): Open label single arm study of CER-001
  Interventions: Drug: CER-001

INTERVENTIONS:
Drug: CER-001 — Weekly injection

SUMMARY:
Despite the availability of several classes of very effective drugs available to treat heterozygous Familial Hypercholesterolemia (HeFH), there remains a large unmet medical need for new, effective and well tolerated therapies. There are a number of therapies given on a chronic basis to reduce long term risk, such as statins, fibrates, niacin, omega 3 fatty acids, resins, cholesterol absorption inhibitors and antiplatelet or anticoagulant drugs, but subjects with heterozygous Familial Hypercholesterolemia remain at high risk for cardiovascular events. There is still a need for acute therapies that can lead to rapid pacification of unstable plaque in order to reduce the risk of these events. This study will assess the effects of CER-001 , a recombinant human Apo-A-1 based HDL mimetic, on indices of atherosclerotic plaque progression and regression as assessed by 3Tesla MRI (3TMRI)and intravascular ultrasound (IVUS) evaluations in patients with HeFH.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female subjects at least 18 years old
* Subject presents heterozygous FH, known CHD and receiving maximally tolerated lipid modifying therapy, at stable doses for at least 3 months
* LDL-C of > 110 mg/dl
* Angiographic evidence of coronary artery disease with suitable "target" coronary artery for IVUS

Exclusion Criteria:

* Confirmed diagnosis of homozygous FH
* Significant health problems (other than cardiovascular disease) in the recent past including blood disorders, cancer, or digestive problems
* Female subjects not meeting the study definition of non child-bearing potential
* Use of an investigational agent within 30 days of the first CER-001 dose
* Receiving current lipid apheresis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in Total Plaque Volume | Baseline and 3 weeks post final dose
  Nominal change in total plaque volume (ACTPV), as assessed by 3D IVUS, from the baseline measurement to the follow-up taken ~3 weeks following the final dose of study medication (approximately 10 weeks after the baseline assessment)

SECONDARY OUTCOMES:
Percent Change in Plaque Volume | Baseline and 3 weeks post final dose
  Percent change in total plaque volume (PCTPV), as assessed by IVUS, from the baseline measurement to the follow up taken approximately 3 weeks following the final dose of study medication (approximately 10 weeks after the baseline assessment)
Change in carotid plaque volume | Baseline and 3 weeks post final dose
  Percent change in total carotid plaque volume, as assessed by 3TMRI, from the baseline measurement to the follow up taken approximately 3 weeks following the final dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Eriksson M, Carlson LA, Miettinen TA, Angelin B. Stimulation of fecal steroid excretion after infusion of recombinant proapolipoprotein A-I. Potential reverse cholesterol transport in humans. Circulation. 1999 Aug 10;100(6):594-8. doi: 10.1161/01.cir.100.6.594. PMID 10441095
- [Background] Nanjee MN, Doran JE, Lerch PG, Miller NE. Acute effects of intravenous infusion of ApoA1/phosphatidylcholine discs on plasma lipoproteins in humans. Arterioscler Thromb Vasc Biol. 1999 Apr;19(4):979-89. doi: 10.1161/01.atv.19.4.979. PMID 10195926
- [Background] Spieker LE, Sudano I, Hurlimann D, Lerch PG, Lang MG, Binggeli C, Corti R, Ruschitzka F, Luscher TF, Noll G. High-density lipoprotein restores endothelial function in hypercholesterolemic men. Circulation. 2002 Mar 26;105(12):1399-402. doi: 10.1161/01.cir.0000013424.28206.8f. PMID 11914243
- [Background] Nieuwdorp M, Vergeer M, Bisoendial RJ, op 't Roodt J, Levels H, Birjmohun RS, Kuivenhoven JA, Basser R, Rabelink TJ, Kastelein JJ, Stroes ES. Reconstituted HDL infusion restores endothelial function in patients with type 2 diabetes mellitus. Diabetologia. 2008 Jun;51(6):1081-4. doi: 10.1007/s00125-008-0975-2. Epub 2008 Apr 4. No abstract available. PMID 18389214
- [Background] Shaw JA, Bobik A, Murphy A, Kanellakis P, Blombery P, Mukhamedova N, Woollard K, Lyon S, Sviridov D, Dart AM. Infusion of reconstituted high-density lipoprotein leads to acute changes in human atherosclerotic plaque. Circ Res. 2008 Nov 7;103(10):1084-91. doi: 10.1161/CIRCRESAHA.108.182063. Epub 2008 Oct 2. PMID 18832751
- [Background] Nissen SE, Tsunoda T, Tuzcu EM, Schoenhagen P, Cooper CJ, Yasin M, Eaton GM, Lauer MA, Sheldon WS, Grines CL, Halpern S, Crowe T, Blankenship JC, Kerensky R. Effect of recombinant ApoA-I Milano on coronary atherosclerosis in patients with acute coronary syndromes: a randomized controlled trial. JAMA. 2003 Nov 5;290(17):2292-300. doi: 10.1001/jama.290.17.2292. PMID 14600188
- [Background] Tardif JC, Gregoire J, L'Allier PL, Ibrahim R, Lesperance J, Heinonen TM, Kouz S, Berry C, Basser R, Lavoie MA, Guertin MC, Rodes-Cabau J; Effect of rHDL on Atherosclerosis-Safety and Efficacy (ERASE) Investigators. Effects of reconstituted high-density lipoprotein infusions on coronary atherosclerosis: a randomized controlled trial. JAMA. 2007 Apr 18;297(15):1675-82. doi: 10.1001/jama.297.15.jpc70004. Epub 2007 Mar 26. PMID 17387133
- [Background] Waksman R, Torguson R, Kent KM, Pichard AD, Suddath WO, Satler LF, Martin BD, Perlman TJ, Maltais JA, Weissman NJ, Fitzgerald PJ, Brewer HB Jr. A first-in-man, randomized, placebo-controlled study to evaluate the safety and feasibility of autologous delipidated high-density lipoprotein plasma infusions in patients with acute coronary syndrome. J Am Coll Cardiol. 2010 Jun 15;55(24):2727-35. doi: 10.1016/j.jacc.2009.12.067. PMID 20538165